CLINICAL TRIAL: NCT01028573
Title: A Randomized, Controlled, Single-Blind Study Comparing the Efficacy, Tolerability and Safety of PEG-3350 (Miralax) and Gatorade With PEG-ELS (Golytely) for Bowel Preparation Prior to Colonoscopy
Brief Title: A Study Comparing PEG-3350 (Miralax) and Gatorade With PEG-ELS (Golytely) for Bowel Preparation Prior to Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: M. Mazen Jamal, MD, VA Long Beach Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 976
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Bowel Preparation for Colonoscopy
Keywords: bowel preparation; colonoscopy
MeSH Terms: interventions — Golytely; gatorade; polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Active Comparator): 4L of PEG-ELS (Golytely) consumed on the evening before colonoscopy
  Interventions: Drug: PEG-ELS (Golytely)
- Group 2 (Experimental): 2L of PEG-ELS (Golytely) consumed on the evening before and 2L consumed on the morning of colonoscopy
  Interventions: Drug: PEG-ELS (Golytely)
- Group 3 (Experimental): 238g of PEG-3350 mixed with 2L of Gatorade
  Interventions: Drug: Miralax mixed with Gatorade
- Group 4 (Experimental): 1L of PEG-3350 + Gatorade
  Interventions: Drug: Miralax

INTERVENTIONS:
Drug: PEG-ELS (Golytely) — 4L consumed evening before colonoscopy
  Arms: Group 1
Drug: PEG-ELS (Golytely) — 2L consumed on the evening before and 2L consumed on the morning of Colonoscopy
  Arms: Group 2
Drug: Miralax mixed with Gatorade — 238g of PEG-3350 (Miralax) mixed with 2L of Gatorade consumed on the evening before colonoscopy
  Arms: Group 3
Drug: Miralax — 1L of PEG-3350 + Gatorade consumed on the evening before and 1L of PEG-3350 + Gatorade consumed on the morning of Colonoscopy
  Arms: Group 4

SUMMARY:
The purpose of this study to to see how well Miralax (PEG-3350) and Gatorade cleans the colon before a colonoscopy and how easy it is to take compared to Golytely (PEG-ELS) bowel preparation solution. Another purpose is to see if taking half of the bowel preparation solution on the evening before the colonoscopy and half on the morning of the colonoscopy will result in a cleaner colon than taking all of the bowel preparation solution on the evening before.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years in age
* Undergoing full colonoscopy for colorectal cancer screening or colon polyp/cancer surveillance or other diagnostic purpose

Exclusion Criteria:

* Allergic to polyethylene glycol
* Pregnant or lactating
* Baseline abnormalities of relevant serum electrolytes including Sodium, Potassium, Calcium, Magnesium and phosphorus
* Congestive Heart Failure NY Heart Assn, Grades III and IV
* Liver Cirrhosis Childs Pugh Class B or C
* Serum Creatinine greater than 1.5
* Previous alimentary tract surgery
* Ongoing symptoms of abdominal pain, bloating, nausea or constipation
* Ileus, suspected bowel obstruction, toxic colitis or megacolon, severe ulcerative colitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Quality of bowel prepreparation/cleanliness scored using the Boston Bowel Preparation Scale | two years

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Jamal, MD, Principal Investigator — VA Long Beach Healthcare System
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States